CLINICAL TRIAL: NCT01588938
Title: External Immobilization Compared to Limited Immobilization Using a Novel Real-time Localization System of the Prostate
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: U.S. Army Medical Research Acquisition Activity (U.S. Federal Agency)
Collaborators: The Geneva Foundation (Other)
Responsible Party: Principal Investigator, Dusten Macdonald, MD, MD, MC, Madigan Army Medical Center
Other Study IDs: W81XWH-08-2-0174, A-15214.1b; W81XWH-08-2-0174 (Other Grant/Funding Number: US Army Medical Research Acquisition Activity); 209099 (Other: Madigan Army IRB)
Record Dates: First submitted 2012-04-26; First posted 2012-05-01 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Prostate Cancer
Keywords: radiation therapy; Calypso
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This prospective study at MAMC evaluates the utility of a rigid pelvic external immobilization compared to limited immobilization using a novel real-time localization system of the prostate. The sample population will include patients referred to the radiation oncology services of both facilities for definitive treatment of prostate cancer. The study will enroll 20 subjects from MAMC and evaluate data on 860 radiation therapy fractions.

Subjects will have Beacon® Transponders implanted into the prostate to more precisely localize the position of the organ during radiation therapy. They will be randomized to rigid pelvic immobilization using a Vac-Lok® system or limited immobilization with a band around the patient's feet. They will then undergo radiation therapy planning with standard planning target margins. The Calypso® 4D Localization System will monitor, in real time, the position of the prostate target and adjust radiation treatments as required to ensure accurate treatment of the prostate gland. The time of, the number, and extent of adjustments will be recorded for analysis.

Hypothesis: 1. When treating only the prostate, treatment with rigid pelvic immobilization is not necessary when using real-time, state-of-the-art motion tracking of the prostate.

DETAILED DESCRIPTION:
Medical application: This study will seek to determine the utility of rigid external pelvic immobilization in patients who are set up using real-time, state-of-the-art motion tracking of the prostate. External immobilization devices have been criticized for being expensive, uncomfortable, time-consuming to make, occupying a lot of space in the treatment area, creating difficulties at the time of CT simulation, challenging for obese patients and obscuring skin marks that can help confirm patient set up. Omitting these devices (if found to be unnecessary) would potentially decrease treatment costs, improve patient comfort during treatment, and reduce overall treatment time. In high risk patients, gaining a better understanding of lymph node positioning relative to Calypso immobilization may allow for decreased PTV margins and therefore decreased normal tissue irradiated during radiation therapy.

Objective(s) of the investigation: This study will look at the efficacy of external pelvic immobilization in definitive radiation therapy of prostate cancer using a unique organ tracking system.

A. Primary Objective: To determine if rigid external pelvic immobilization demonstrates a reduction in positioning errors. This will be assessed by determining the median, mean and range of shifts performed in all 3 dimensions as part of initial isocenter set-up and during treatment using the Calypso system.

B. Secondary Objectives: The study will determine the simulation time, set up time, treatment time, total time and number of treatment interventions (repositioning/pausing) caused by organ/target motion beyond planning target volume (PTV) margin using real time localization. In the subset of high-risk patients, this study will assess positioning of the lymph node target using the combination of rigid external pelvic immobilization and the Calypso system.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate
* Stage T1 -T3a, N0 or NX, M0
* Ability to comply with study schedule
* Age 40 or older
* Zubrod PS 0 or 1 (appendix 1)
* Signed informed consent

Exclusion Criteria:

* Node positive or metastatic prostate cancer
* Prior treatment of prostate cancer with surgery, chemotherapy, cryotherapy or brachytherapy
* History of prior pelvic radiotherapy
* History of abdominoperineal resection
* History of inflammatory bowel disease or connective tissue disease
* History of HIV infection
* History of chronic prostatitis or chronic cystitis
* History of bleeding disorder or any active anticoagulation (excluding ASA) which cannot be safely discontinued for beacon placement
* PT or INR outside normal range for institution
* Active implanted devices such as cardiac pacemakers and automatic defibrillators.
* Prosthetic implants in the pelvic region that contain metal or conductive materials (eg., an artificial hip).
* Patients with maximum anterior-posterior separation through the torso minus the height of the center of the prostate greater than 17 cm (technical reason for Calypso System, see appendix 5).

Min Age: 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will include patients with prostate cancer for whom definitive radiation therapy is planned to the prostate. Patients will be referred from Urology and Radiation Oncology.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2009-12; Primary Completion 2016-09 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Rigid external pelvic immobilization demonstrates a reduction in positioning errors. | Measured at every treatment fraction for a total of approximately 8.5 weeks
  This will be assessed by determining the median, mean and range of shifts performed in all 3 dimensions as part of initial isocenter set-up and during treatment using the Calypso system.

SECONDARY OUTCOMES:
Simulation time, set up time, treatment time, total time and number of treatment interventions (repositioning/pausing) caused by organ/target motion beyond planning target volume (PTV) margin using real time localization. | Measured at simluation and every treatment fraction for a total of approximately 10 weeks
  During each radiation treatment fraction, therapists will record these timepoints and number/duaration of treatment inverventions.
Positioning of the lymph node target using the combination of rigid external pelvic immobilization and the Calypso system. | Measured at every treatment fraction for a total of approximately 8.5 weeks
  This will be analyzed in the subset of high-risk patients.

CONTACTS AND LOCATIONS:
Overall Officials: Dusten Macdonald, MD, Principal Investigator — Department of the Army
Locations (1):
- Madigan Healthcare System, Tacoma, Washington, United States